CLINICAL TRIAL: NCT00688181
Title: The Prefyx PPS™ System eRegistry
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: U8043
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Results first posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects treated with the Prefyx PPS System: All patients presenting to the institution for treatment of female Stress Urinary Incontinence (SUI), excluding those patients meeting any of the contraindications as noted in the Directions For Use.
  Interventions: Device: The Prefyx PPS™ Pre-pubic Sling System

INTERVENTIONS:
Device: The Prefyx PPS™ Pre-pubic Sling System — device designed to treat female stress urinary incontinence (SUI).

SUMMARY:
Registry to gather information about the long term use of the Prefyx PPS System for the treatment of Stress Urinary Incontinence (SUI).

DETAILED DESCRIPTION:
Registry to gather information about the long term use of the Prefyx PPS System which utilizes a pre-pubic surgical approach (device is to be placed in front of the pubic bone) for the treatment of SUI. No additional procedures are required beyond the physician's standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for treatment of female Urinary Stress Incontinence (SUI)

Exclusion Criteria:

* Pregnant patients, patients with the potential for future growth or patients that are considering future pregnancies.
* Any patients with soft tissue pathology into which the implant is to be placed.
* Patients with any pathology which would compromise implant placement.
* Patients with any pathology, such as blood supply limitations or infections that would compromise healing.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients presenting to the institution for treatment of female Urinary Stress Incontinence (SUI) should be eligible for enrollment in the PPS eRegistry. However, any patient meeting any of the contraindications should NOT be included as noted in the Directions For Use. Minors are excluded from the registry per contraindications in which mesh implants are contraindicated in 'patients with the potential for future growth'.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Walsh, M.D., Study Director — Boston Scientific Corporation
Locations (5):
- United States (5):
  - South Florida Urology Center, Pembroke Pines, Florida
  - OB/GYN Specialists of the Palm Beaches, West Palm Beach, Florida
  - Urology Specialists of Atlanta, LLC /Northside Hospital, Atlanta, Georgia
  - Affiliates in Urology, Westland, Michigan
  - HillCrest Medical Center, Tulsa, Oklahoma

REFERENCES:
- See also: Related Info — http://www.Prefyx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 58 patients were enrolled at 5 centers in the United States from November 2006 to November 2008. However, only 36 patients' data are included in this final synopsis report. A total of 22 patients were removed from the study database due to informed consent form non-compliance.
Groups:
- Subjects Treated With the Prefyx PPS System: All patients presenting to the institution for treatment of female Stress Urinary Incontinence (SUI) and treated using the Prefyx PPS System, excluding those patients meeting any of the contraindications as noted in the Directions For Use.
Period: Overall Study
Arm/Group | Subjects Treated With the Prefyx PPS System
Started | 36
Completed | 13
Not Completed | 23
Not completed — Lost to Follow-up | 17
Not completed — Unknown Reason | 4
Not completed — Non-clinical Reason | 2

BASELINE CHARACTERISTICS:
Groups:
- Subjects Treated With the Prefyx PPS System: All patients presenting to the institution for treatment of female Urinary Stress Incontinence (SUI) and treated with the Prefyx PPS System, excluding those patients meeting any of the contraindications as noted in the Directions For Use.
Arm/Group | Subjects Treated With the Prefyx PPS System
Number analyzed (Participants) | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (13.8)
Age, Customized [Mean (Full Range); unit: years]
  Age Range in Years | 60.4 [34 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Remain Continent or Improved Following Treatment Through 3 Months Follow-up
Description: Continence was measured by participant subjective feedback. Responses included: cured, significantly improved, slightly improved, same, slightly worse, or significantly worse
Time Frame: 3 months
Population: 26 patients analyzed at 3 months
Measure: Number; unit: Participants
Groups:
- Subjects Treated With the Prefyx PPS System: All patients presenting to the institution for treatment of female Stress Urinary Incontinence (SUI) and treated with the Prefyx PPS System, excluding those patients meeting any of the contraindications as noted in the Directions For Use.
Arm/Group | Subjects Treated With the Prefyx PPS System
Number analyzed (Participants) | 26
Participants | 26

2. Primary Outcome: Number of Participants Who Remain Continent or Improved Following Treatment Through 12 Months Follow-up
Description: as for outcome 1
Time Frame: 12 months
Population: 12 patients analyzed at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Subjects Treated With the Prefyx PPS System
Number analyzed (Participants) | 12
Participants | 8

3. Primary Outcome: Number of Participants Who Report Substantial Improvement and Consider the Surgery Successful, as Measured by the Patient's Global Impression
Description: Substantial improvement is measured by the participants' subjective feedback of their incontinence if they are cured, improved, same, or worse. Patients' Global Impression measures satisfaction (satisfied, or not satisfied).
Time Frame: 12 months
Population: 11 completed the Global Impression at 12 months
Measure: Number; unit: Participants
Groups:
- Subjects Treated With the Prefyx PPS System: All patients presenting to the institution for treatment of female Urinary Stress Incontinence (SUI), excluding those patients meeting any of the contraindications as noted in the Directions For Use.
Arm/Group | Subjects Treated With the Prefyx PPS System
Number analyzed (Participants) | 11
Participants | 7

4. Primary Outcome: Number of Participants With Adverse Events
Description: Adverse events were collected throughout the study and tabulated per severity, seriousness, and device-relatedness.
Time Frame: 12 months
Population: Analysis was per protocol
Measure: Number; unit: Participants
Arm/Group | Subjects Treated With the Prefyx PPS System
Number analyzed (Participants) | 36
Participants | 23

ADVERSE EVENTS:
Arm/Group | Subjects Treated With the Prefyx PPS System
Serious Adverse Events (participants affected / at risk) | 19/36
Other Adverse Events (participants affected / at risk) | 13/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Treated With the Prefyx PPS System (N=36)
Atrophy, Moderate (Reproductive system and breast disorders) | 1 (1)
Erosion, Moderate (Reproductive system and breast disorders) | 1 (1)
Incontinence, Mild (Renal and urinary disorders) | 6 (6)
Incontinence, Moderate (Renal and urinary disorders) | 4 (4)
Infection, Mild (Infections and infestations) | 2 (2)
Infection, Moderate (Infections and infestations) | 1 (1)
Nausea, Moderate (Gastrointestinal disorders) | 1 (1)
Numbness, Mild (Nervous system disorders) | 1 (1)
Other, Mild (General disorders) | 1 (1)
Other, Moderate (General disorders) | 1 (1)
Pain, Mild (Nervous system disorders) | 4 (4)
Pain, Severe (Nervous system disorders) | 1 (1)
Restlessness, Moderate (Nervous system disorders) | 1 (1)
Vaginal Burning, Moderate (Reproductive system and breast disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects Treated With the Prefyx PPS System (N=36)
Atrophy, Moderate (Reproductive system and breast disorders) | 1 (1)
Bleeding, Mild (General disorders) | 2 (2)
Difficulty Breathing, Mild (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hematoma, Mild (Skin and subcutaneous tissue disorders) | 1 (1)
Hematuria, Mild (Renal and urinary disorders) | 1 (1)
Incontinence, Moderate (Renal and urinary disorders) | 1 (1)
Other, Mild (General disorders) | 1 (1)
Pain, Mild (Nervous system disorders) | 3 (3)
Pain, Moderate (Nervous system disorders) | 1 (1)
Vomitting, Moderate (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No